CLINICAL TRIAL: NCT01600417
Title: Radiologic Presentation of Lumbo-sacral Instability Using a Custom Made Table - a Pilot Study
Brief Title: Investigation of Lumbo-sacral Instability Using Custom Made Table - a Pilot Study
Status: Terminated | Type: Observational
Why Stopped: principal investigator has left the institution
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2011-11
Record Dates: First submitted 2012-05-08; First posted 2012-05-17 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Low Back Pain
Keywords: low back pain; spine; lumbar spine; lumbar instability; radiology; functional radiology
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- clinical suspicion of lumbar instability

SUMMARY:
The aim of the study is to evaluate the feasibility and validity of conventional radiographs of the lumbo-sacral spine when the patient is lying on a special table which facilitates maximal lumbo-sacral flexion. The results gained from the radiographs with the patient on the table will be compared with those gained from standard flexion-extension radiographs of the lumbo-sacral spine.

DETAILED DESCRIPTION:
After enrollment in the study patients will complete a set of questionnaire concerning degree, extent and quality of their low back problem. Afterwards a lateral conventional radiograph of the lumbar spine with the patient on a custom made positioning table will be taken. The table facilitates optimal flexion of the lumbar spine. Afterwards sagittal translation and rotation are measured on the flexion-extension radiographs and the radiograph taken on the custom made table. Differences between the measurements will be determined.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain (≥ 3 months)
* clinical suspicion of lumbo-sacral instability
* functional conventional radiographs of lumbar spine
* pain intensity > 4 / 10 on visual analogue scale
* age 20-60 years

Exclusion Criteria:

* radicular pain
* pain at more than two locations
* lumbar spine surgery
* scoliosis
* lumbar spondylolysis
* lumbar spondylodiscitis
* anatomic aberrations of lumbar spine
* unconsolidated spine fractures
* neurologic deficits
* spine tumor
* neuromuscular disease
* rheumatic disease
* severe osteoporosis
* radiotherapy within the last 5 years
* pregnancy
* insufficient German language skills
* no informed consent

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients suffering from chronic low back pain and clinical suspicion of lumbar instability.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
sagittal translation | baseline
  sagittal translation of L1-L5 on conventional radiographs

SECONDARY OUTCOMES:
patient characteristics | baseline
  age
SF-36 questionnaire | baseline
visual analogue scale of low back pain | baseline
Short Form McGill questionnaire | baseline
sagittal rotation | baseline
  sagittal rotation of L1-L5 on conventional radiographs
Oswestry questionnaire | baseline
patient characteristics | baseline
  weight
patient characteristics | baseline
  height

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus Aebli, Prof, Principal Investigator — Swiss Paraplegic Centre
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland